CLINICAL TRIAL: NCT02099643
Title: Crucial Areas on Atrial Fibrillation Termination by Substrate Ablation: Relevance to Anatomy
Brief Title: Crucial Areas on AF Termination
Status: Completed | Type: Observational
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Principal Investigator, SEITZ JULIEN, CARDIOLOGIST, Hospital St. Joseph, Marseille, France
Other Study IDs: HSJ-2013-03
Record Dates: First submitted 2014-03-26; First posted 2014-03-31 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Atrial Fibrilation Termination Endpoint

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
Recent data has demonstrated that focal sources are determinant in human atrial fibrillation (AF) perpetuation.

The investigators sought to identify crucial areas for AF perpetuation during our routine electrogram (EGM)-based substrate ablation.

ELIGIBILITY:
Inclusion Criteria:

* Atrial Fibrilation
* Undergoing EGM-based substrate ablation

Exclusion Criteria:

* Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with symptomatic Atrial Fibrilation undergoing EGM-based substrate ablation were included.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2008-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Atria fibrillation termination during procedure | 240 min
  conversion to atrial tachycardia (AT) or sinus rhythm

SECONDARY OUTCOMES:
Crucial points | 240 min
  Crucial points were defined by areas where ablation immediately extended the cycle length> 20% of AF CL, or regularized Atrial Fibrilation (AF) into Atrial Tachycardia (AT) or converted AF (or AT) into Sinus Rythm

CONTACTS AND LOCATIONS:
Locations (4):
- France (3):
  - Hopital Saint Joseph, Marseille
  - Hôpital Privé Jacques Cartier;, Massy
  - Institut Mutualiste Montsouris;, Paris
- Morphology Unit Royal Brompton Hospital, London, United Kingdom